CLINICAL TRIAL: NCT02838433
Title: Study of Anti-telomerase T CD4 Immunity in Melanoma: Predictive Biomarker and Implications for Immunotherapy
Brief Title: Study of Anti-telomerase T CD4 Immunity in Melanoma
Acronym: LyTéloMel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: T/2011/03
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological samples (Experimental): Blood samples will be collected :
  * at baseline,
  * 6 months after the first-line therapy or at disease progression (if occurs first).
  In particular case of patient with immunotherapy or targeted therapy, 3 blood samples will be collected :
  * at baseline
  * 3 months after the initiation of immunotherapy or targeted therapy
  * at disease progression Tumor tissues will be collected if available.
  Interventions: Other: biological samples

INTERVENTIONS:
Other: biological samples — blood and tissue samples

SUMMARY:
The impressive clinical responses obtained with immune checkpoint inhibitors (anti-PD-1/PDL-1, anti-CTLA-4) indicate that the presence of preexisting antitumor immune response might be required for their efficacy and highlight the critical role of antitumor T cell immunity.

Recent progresses on the field of tumor immunology underline the critical role of CD4 helper 1 T lymphocyte (TH1) in the control of innate and adaptive anticancer immunity. Therefore, monitoring tumor specific TH1 response could be relevant in cancer patients.

In order to monitor tumor-specific CD4 Th1 responses in most cancer patients, the investigators team have previously described novel promiscuous peptides (referred as UCP: Universal Cancer Peptides) derived from human telomerase (TERT), a prototype of shared tumor antigen.

By using UCP-based immuno-assay, UCP specific Th1 immune responses will be evaluated in this study in melanoma before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient with melanoma, any stade, without history of anti-cancer treatment (surgery, chemotherapy, targeted therapy, immunotherapy...) except for patients with stade IV melanoma for which immunotherapy or targeted therapy is considered. In this case, a first-line chemotherapy treatment is allowed
* written informed consent

Exclusion Criteria:

* patient with immunosuppressive treatment
* active autoimmune diseases, HIV, hepatitis C or B virus
* patients under guardianship, curatorship or under the protection of justice, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Presence of spontaneous UCP-specific Th1 responses measured by ELISPOT assay | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Besançon, Besançon, France